CLINICAL TRIAL: NCT03829488
Title: An Investigator-initiated, Pragmatic, Registry-based, Multi-centre, Double-blind, Randomised Controlled Trial Evaluating the Effect of Plasmalyte Versus 0.9% Saline on Early Kidney Transplant Function in Deceased Donor Kidney Transplantation
Brief Title: Better Evidence for Selecting Transplant Fluids
Acronym: BEST-Fluids
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Australian Government Department of Health and Ageing (Other Government); Health Research Council, New Zealand (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AKTN 15.02; ACTRN12617000358347 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2019-01-21; First posted 2019-02-04 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2021-09

CONDITIONS: End Stage Kidney Disease; Delayed Graft Function; Kidney Transplant; Complications
MeSH Terms: conditions — Kidney Failure, Chronic; Delayed Graft Function | interventions — Plasma-lyte 148; Infusions, Intravenous; Plasmalyte A; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma-Lyte 148 (approx. pH 7.4) IV Infusion (Experimental): Plasma-Lyte 148 (approx. pH 7.4) IV Infusion intravenous fluid therapy will be used for all maintenance, replacement and resuscitation purposes from randomization onwards until 48 hours post-transplant, or until fluid therapy is no longer required, if earlier.
  Interventions: Drug: Plasma-Lyte 148 (approx. pH 7.4) IV Infusion
- 0.9% SODIUM CHLORIDE 9g/L injection BP (Active Comparator): 0.9% saline intravenous fluid therapy will be used for all maintenance, replacement and resuscitation purposes from randomization onwards until 48 hours post-transplant, or until fluid therapy is no longer required, if earlier.
  Interventions: Drug: 0.9% SODIUM CHLORIDE 9g/L injection BP

INTERVENTIONS:
Drug: Plasma-Lyte 148 (approx. pH 7.4) IV Infusion — Plasma-Lyte 148 (approx. pH 7.4) IV Infusion is a sterile, clear, non-pyrogenic isotonic solution and when administered intravenously is a source of water, electrolytes and calories. Plasma-Lyte 148 intravenous infusion is indicated as a source of water & electrolytes or as an alkalinising agent.
  Other Names: Plasma-Lyte 148®; Plasmalyte; Balanced crystalloid solution
  Arms: Plasma-Lyte 148 (approx. pH 7.4) IV Infusion
Drug: 0.9% SODIUM CHLORIDE 9g/L injection BP — Sodium chloride (0.9% saline) infusion is a sterile, non-pyrogenic solution of sodium chloride in Water for Injections. The concentration of sodium chloride is 154mmol/L. Sodium chloride (0.9%) intravenous infusion is indicated for extra-cellular fluid replacement and in the management of metabolic alkalosis in the presence of fluid loss, and for restoring or maintaining the concentration of sodium and chloride ions.
  Other Names: 0.9% saline; Normal saline; Isotonic saline
  Arms: 0.9% SODIUM CHLORIDE 9g/L injection BP

SUMMARY:
End-stage kidney disease (ESKD) is a significant, expensive health problem. Kidney transplantation improves survival, quality of life, and is much cheaper than dialysis treatment for ESKD. However sometimes kidney transplants from a deceased donor function poorly after surgery, and a period of continued dialysis is needed, a condition known as delayed graft function (DGF). In addition to complicating recovery, DGF can adversely affect long-term kidney function and the health of the recipient.

Intravenous fluids given during and after transplantation (usually 0.9% sodium chloride or saline) are critical to preserve kidney transplant function, but there is evidence that 0.9% saline may not be the safest fluid to use due to its high chloride content.

BEST Fluids is a randomised controlled trial that aims to find out whether using a balanced low-chloride solution - Plasma-Lyte 148® - as an alternative to normal saline in deceased donor kidney transplantation, will improve kidney transplant function, reduce the impact of DGF, and improve long-term outcomes for patients.

DETAILED DESCRIPTION:
End-stage kidney disease is a significant public health problem worldwide, and its treatment imposes a high healthcare burden and cost. Kidney transplantation is considered the best treatment for ESKD, offering improved survival and quality of life at significantly lower cost that dialysis. However, many kidney transplants fail prematurely due in part due to injury sustained at the time of transplantation. Delayed graft function (DGF), i.e. the requirement for dialysis early after transplantation, affects approximately 30% of deceased donor kidney transplants, and increases the risk of graft failure and mortality.

Intravenous fluids are a critical, albeit inexpensive, aspect of care that impacts early transplant function with normal (0.9%) saline the current standard care at most centres. However, normal saline may in fact be harmful in the setting of kidney transplantation due to its high chloride content relative to plasma, causing metabolic acidosis, acute kidney injury and thus potentially increasing the risk of DGF. Utilising a balanced low-chloride crystalloid solution such as Plasma-Lyte 148® (Plasmalyte) as an alternative to 0.9% saline may therefore improve outcomes after kidney transplantation.

The BEST-Fluids study is an investigator-initiated, pragmatic, registry-based, multi-centre, double -blind randomised, controlled trial. The primary objective of the study is to evaluate the effect in deceased donor kidney transplant recipients of intravenous therapy with Plasmalyte versus 0.9% saline, commencing pre-operatively and continuing until intravenous fluids are no longer required or 48 hours post-transplant (whichever is earliest), on DGF, defined as the requirement for dialysis in the first seven days post-transplant.

Patients admitted for a deceased donor kidney transplant at participating centres will be invited to participate in the study prior to transplant surgery. Following informed consent, participants will be randomised to receive either blinded Plasmalyte or blinded 0.9% saline for all intravenous fluid therapy purposes until 48 hours post-transplant. The volume and rate of fluid therapy will be determined by treating clinicians; all other treatments will be as per local standard of care. Participants will be enrolled, randomised and followed up using ANZDATA, the Australia & New Zealand Dialysis & Transplant Registry.

The trial was prospectively registered with Australia New Zealand Clinical Trials Registry (ANZCTR) on 08/03/2017 (ACTRN12617000358347).

ELIGIBILITY:
Inclusion Criteria:

1. Adult or child with End-Stage Kidney Disease, of any cause, on maintenance dialysis, or who has pre-dialysis stage 5 chronic kidney disease with an estimated Glomerular Filtration Rate of <15 mL/min/1.73m2, AND
2. Planned deceased donor kidney transplant from a brain-death (DBD) or circulatory-death (DCD) organ donor within 24 hours, AND
3. Written informed consent, or consent given by their parent or guardian (if age <18), or other authorised person

Exclusion Criteria:

1. Planned live donor kidney transplant (except where this is cancelled in favour or transplantation from a deceased donor)
2. Planned multi-organ transplant (dual or en-bloc kidney transplants are not excluded)
3. Children of weight <20 kg, or a child that the treating physician believes should not be included in a study of blinded fluids due to their small body size
4. Known hypersensitivity to the trial fluid preparations or packaging

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 808 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
The proportion of participants with Delayed Graft Function | 7 Days
  Delayed Graft Function defined as receiving treatment with any form of dialysis in the first seven days after transplant

SECONDARY OUTCOMES:
Early Kidney Transplant Function | a. Duration of Delayed Graft Function - 12 Weeks; b. Rate of recovery of kidney transplant graft function - 2 Days
  Early Kidney Transplant Function, a ranked composite of
  1. Duration of Delayed Graft Function Description: Participants who require dialysis within seven days post-transplant, the time from transplant to the final dialysis treatment in days (up to 84 days/12 weeks) will be ranked from best to worst (longer times are worse).
  2. Rate of recovery of kidney transplant graft function Description: for participants who do not require dialysis, graft function assessed using the creatinine reduction ratio on post-transplant day two (CRR2) will be ranked from best to worst (smaller reductions are worse).
Number of dialysis sessions | First 28 days post-transplant
  The number of dialysis sessions
Total duration of dialysis | 12 Weeks
  The total duration of dialysis in days
Creatinine reduction ratio from day 1 to day 2 post-transplant | Day 1 to Day 2 post-transplant
  Creatinine reduction ratio from day one to day two measured using serum assay, for those who do not require dialysis within the first 7 days
Reduction in serum creatinine of greater than or equal to 10% | First 7 days post-transplant
  The proportion of subjects with a reduction in serum creatinine of greater than or equal to 10% on three consecutive days in the first 7 days post-transplant
Serum creatinine trends over 52 weeks | 12 months
  Serum creatinine trends measured over 52 weeks
Incidence of serum potassium greater than or equal to 5.5 mmol/L | First 48 hours post-transplant
  Serum potassium greater than or equal to 5.5 mmol/L measured by serum assay
Peak potassium level | First 48 hours post-transplant
  Peak potassium level, measured by serum assay
Treatment for hyperkalaemia | First 48 hours post-transplant
  Treatment for hyperkalaemia with dialysis, Ca2+-gluconate, insulin, beta-agonists, sodium bicarbonate or ion exchange resins in the first 48 hours post-transplant
Incidence of significant fluid overload | Baseline to day 2
  Incidence of significant fluid overload defined as >5% weight gain
Aggregate urine output | Until day 2 post-transplant
  Aggregate urine output until day 2 post-transplant
Requirement for inotropic support (use of vasopressors or other drugs to maintain adequate blood pressure) | Intra- and post-operatively to Day 2
  Requirement for inotropic support both intra- and post-operatively to Day 2
Number of acute rejection episodes | 12 months
  Number of acute rejection episodes in the first 52 weeks as reported by ANZDATA routine data capture and as assessed by treating physicians
Number of renal transplant biopsies | First 28 days post-transplant
  Number of renal transplant biopsies performed in the first 28 days post-transplant
Death from all causes | Up to 52 weeks
  Death from all causes up to 52 weeks
Graft survival | 12 months
  Graft survival and death-censored graft survival as reported by ANZDATA and assessed by treating physician
Graft function | 4, 12, 26 and 52 weeks
  Graft function (estimated glomerular filtration rate; eGFR) at 4, 12, 26 and 52 weeks
Health-related quality of life | Baseline, day 7, day 28, week 12, week 26, and week 52
  Health-related quality of life measured using EuroQol EQ-5D-5L for adults, and EQ-5D-Y in children under 18 years. EQ-5D has descriptive and visual analogue scale (VAS). Descriptive system consists of five dimensions mobility, self-care, usual activities, pain/discomfort and anxiety/depression. VAS records patient's self-rated health on vertical visual analogue scale with endpoints best to worst health with 0 being worst and 100 being best health.
Length of hospital stay | 12 months
  Length of hospital stay over 12 months using linked data state and country based health data
Healthcare resource use | 12 months
  Healthcare resource use over 12 months using linked data state and country based health data
Cost-effectiveness | 12 months
  Cost-effectiveness over 12 months using linked data state and country based health data

CONTACTS AND LOCATIONS:
Overall Officials: Michael Collins, MBChB,FRACP,PhD, Study Chair — Auckland District Health Board & The University of Auckland; Steven Chadban, BMed(hons),FRACP,PhD, Principal Investigator — Sydney Local Health District & The University of Sydney
Locations (18):
- Australia (14):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Queensland Children's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St Vincent's Hospital (Melbourne) Ltd, Melbourne, Victoria
  - Austin Health, Melbourne, Victoria
  - Monash Children's Hospital, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital, Perth, Western Australia
- New Zealand (4):
  - Auckland City Hospital, Auckland
  - Starship Children's Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Wellington Hospital, Wellington

IPD SHARING:
Plan to Share IPD: Yes
Yes Individual participant data that underlie the results reported in the primary publication, after de-identification (text, tables, figures and appendices) will be available for individual participant data meta-analysis.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 2 years and ending 5 years following main publication. Proposals may be submitted up to 5 years following article publication. After 5 years, the data will be available in our University's data warehouse but without investigator support other than deposited metadata.
Access Criteria: An independent review board will assess proposals based on the following criteria: sound science, benefit-risk balancing and research team expertise.

REFERENCES:
- [Derived] Collins MG, Fahim MA, Pascoe EM, Hawley CM, Johnson DW, Varghese J, Hickey LE, Clayton PA, Dansie KB, McConnochie RC, Vergara LA, Kiriwandeniya C, Reidlinger D, Mount PF, Weinberg L, McArthur CJ, Coates PT, Endre ZH, Goodman D, Howard K, Howell M, Jamboti JS, Kanellis J, Laurence JM, Lim WH, McTaggart SJ, O'Connell PJ, Pilmore HL, Wong G, Chadban SJ; BEST-Fluids Investigators; Australasian Kidney Trials Network. Balanced crystalloid solution versus saline in deceased donor kidney transplantation (BEST-Fluids): a pragmatic, double-blind, randomised, controlled trial. Lancet. 2023 Jul 8;402(10396):105-117. doi: 10.1016/S0140-6736(23)00642-6. Epub 2023 Jun 18. PMID 37343576
- [Derived] Pascoe EM, Chadban SJ, Fahim MA, Hawley CM, Johnson DW, Collins MG; BEST-fluids Investigators and the Australasian Kidney Trials Network. Statistical analysis plan for Better Evidence for Selecting Transplant Fluids (BEST-Fluids): a randomised controlled trial of the effect of intravenous fluid therapy with balanced crystalloid versus saline on the incidence of delayed graft function in deceased donor kidney transplantation. Trials. 2022 Jan 18;23(1):52. doi: 10.1186/s13063-021-05989-w. PMID 35042554
- [Derived] Collins MG, Fahim MA, Pascoe EM, Dansie KB, Hawley CM, Clayton PA, Howard K, Johnson DW, McArthur CJ, McConnochie RC, Mount PF, Reidlinger D, Robison L, Varghese J, Vergara LA, Weinberg L, Chadban SJ; BEST-Fluids Investigators and the Australasian Kidney Trials Network. Study Protocol for Better Evidence for Selecting Transplant Fluids (BEST-Fluids): a pragmatic, registry-based, multi-center, double-blind, randomized controlled trial evaluating the effect of intravenous fluid therapy with Plasma-Lyte 148 versus 0.9% saline on delayed graft function in deceased donor kidney transplantation. Trials. 2020 May 25;21(1):428. doi: 10.1186/s13063-020-04359-2. PMID 32450917
- See also: Australasian Kidney Trials Network Website — http://aktn.org.au/best-fluids
- See also: Study protocol paper — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-020-04359-2
- See also: Statistical Analysis Plan paper — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-021-05989-w#change-history
- See also: Baseline characteristics and representativeness paper — https://journals.lww.com/transplantationdirect/Fulltext/2022/12000/Baseline_Characteristics_and_Representativeness_of.5.aspx?context=LatestArticles